CLINICAL TRIAL: NCT04784468
Title: DNA Damage and Oxidative Stress in Hospitalized COVID-19 Patients Compared to Healthy Controls: A Case-control Study
Brief Title: DNA Damage and Oxidative Stress in Hospitalized COVID-19 Patients
Acronym: ABCD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Vienna (Other)
Collaborators: SMZ-Ost Donauspital (Other)
Responsible Party: Principal Investigator, Wagner Karl-Heinz, Professor of Human Nutrition, University of Vienna
Other Study IDs: UNIVIE_Covid_Oxstress
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: DNA damage; Oxidative Stress; Inflammation
MeSH Terms: conditions — COVID-19; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Covid-19: Covid-19 patients
  Interventions: Other: No intervention
- Influenza: Influenza patients
  Interventions: Other: No intervention
- Cotrol: Control group
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Case-control design, one single investigation

SUMMARY:
The severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is responsible for the coronavirus disease 2019 (COVID-19) pandemic challenging health systems worldwide.

While there is a clear correlation between oxidative stress markers and the severity of many viral diseases such as hepatitis C, for SARS-CoV clinical data is limited.

The investigators aim at 1.) investigating DNA damage, oxidative stress, inflammation, and aging markers in COVID-19 patients and compare them with age and gender matched healthy controls and patients with influenza; and 2.) investigating all aforementioned parameters during "cytokine storm" via repeated blood sampling.

ELIGIBILITY:
Covid 19 group:

Inclusion Criteria:

* gender: female/male
* age: ≥40 years
* patients admitted at the emergency department
* COVID-19 suspected patients
* able to give written informed consent

Exclusion Criteria:

* children (≤ 18 years) and adults 19-39 years
* not hospitalized, but confirmed COVID-19 patients (outpatients)
* patients without definitive COVID-19 confirmation

Control group:

Inclusion criteria:

* gender: female/male
* age: ≥40 years
* absence of severe illnesses/serious diseases
* able to give written informed consent

Exclusion criteria:

* children (≤ 18 years) and adults 19-39years
* any current or past clinically significant pathology/disease (comorbidity) such as:

  * Malignancies
  * Cardiovascular diseases
  * Diabetes mellitus (I and II)
  * Obesity class III (BMI >40)
  * Other severe diseases (e.g. renal, hepatic, thyroid disease, bone metabolic diseases, rheumatoid osteoarthritis, human immunodeficiency syndrome, …)

Influenza group:

Inclusion criteria:

* gender: female/male
* age: ≥40 years
* patients admitted at the emergency department
* influenza suspected patients
* able to give written informed consent

Exclusion criteria:

* children (≤ 18 years) and adults 19-39 years
* patients without definitive influenza confirmation

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Covid 19 patients:
  Cases after hospital admission.
  Influenza:
  Cases after confirmed influenza diagnosis
  Healthy controls:
  Healthy subjects from the general population
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
DNA damage | Baseline
  Compare DNA damage (% of DNA in the tail; measured by the comet assay) between hospitalized COVID-19 patients to influenza patients and healthy controls.

SECONDARY OUTCOMES:
The investigators will consider further DNA damage parameter | Baseline
  Compare other DNA damage endpoints measured with the comet assay (i.e. tail length, tail moment and damage index) between hospitalized COVID-19 patients to influenza patients and healthy controls.
The investigators will consider oxidative stress marker | Baseline
  Compare oxidative stress biomarker malondialdehyde, FRAP, GSH, GSSG (all µmol/L) and the ration GSH/GSSG between hospitalized COVID-19 patients to influenza patients and healthy controls.
The investigators will consider inflammatory marker | Baseline
  Compare inflammatory marker Interleukin 1 (IL-1), IL-6, IL-8, IL-10, TNF-alpha (all rfU) and CRP (mg/dl) between hospitalized COVID-19 patients to influenza patients and healthy controls.
The investigators will consider the phenotypic age marker | Baseline
  Compare the phenotypic age marker between hospitalized COVID-19 patients to influenza patients and healthy controls.
The investigators will consider RDA and DNA gene expression | Baseline
  Compare RNA and DNA gene expression between hospitalized COVID-19 patients to influenza patients and healthy controls.
The investigators will consider clinical biochemistry marker | Baseline
  Compare clinical biochemistry (Total cholesterol (mg/dl), LDL-cholesterol (mg/dl), triglycerides (mg/dl), blood glucose (mg/dl), uric acid (mg/dl)) between hospitalized COVID-19 patients to influenza patients and healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik Donaustadt, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided